CLINICAL TRIAL: NCT06206278
Title: A Phase II, Multicenter, Open-Label, Single Arm Study of Oral Infigratinib Monotherapy in Patients With Locally Advanced or Metastatic Gastric Cancer or Gastroesophageal Junction Adenocarcinoma, Who Harboring FGFR2 Gene Amplification
Brief Title: Evaluation of Infigratinib in Patients With Locally Advanced or Metastatic Gastric Cancer or GEJ Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reason
Sponsor: LianBio LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB1001-203
Record Dates: First submitted 2023-11-29; First posted 2024-01-16 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; FGFR2
MeSH Terms: conditions — Stomach Neoplasms | interventions — infigratinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infigratinib (Experimental): Infigratinib 125 mg orally daily, 3 weeks on, 1 week off. . In patients with mild liver function abnormalities or mild renal impairment, the starting dose is 100 mg.
  Interventions: Drug: Infigratinib

INTERVENTIONS:
Drug: Infigratinib — Infigratinib is a selective ATP-competitive inhibitor of fibroblast growth factor receptor (FGFR) 1-3 that inhibits FGFR downstream signaling and proliferation in human cancer cell lines with FGFR genetic alterations, significantly inhibiting the growth of several types of cancers driven by FGFR amplification, fusion and mutation.
  Other Names: BGJ398; BBP-831

SUMMARY:
This is a multicenter, open-label, single arm phase II study to evaluate the efficacy and safety of Infigratinib in patients with locally advanced or metastatic GC or GEJ patient with FGFR2 gene amplification, who have failed at least 2 lines of previous standard systemic treatment .

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Histologically or cytologically confirmed locally advanced or metastatic gastric adenocarcinoma, or gastroesophageal junction adenocarcinoma.
* Failed at least 2 lines of prior systemic therapy
* Willing to undergo tumor biopsy or provide FFPE samples for central lab testing.
* At least one measurable tumor lesion by RECIST v1.1
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1.
* Life expectancy ≥3 months.
* Willing to participate in this study and sign informed consent form, able to read and understand the study, follow the procedures.

Exclusion Criteria:

* History of other primary malignancies within 3 years except adequately treated in situ carcinoma of the cervix or non-melanoma carcinoma of the skin or any other curatively treated malignancy that is not expected to require treatment for recurrence during the study.
* Previous or current treatment of a mitogen-activated protein kinase (MAPK-MEK) or selective FGFR inhibitor.
* Any known hypersensitivity to infigratinib or its excipients.
* History and/or current evidence of extensive tissue calcification.
* Current evidence of endocrine alterations of calcium/phosphate homeostasis.
* Have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral infigratinib (such as, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).14. Laboratory abnormality as defined in protocol.
* Considered unsuitable to participate in the study by Investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Week9/17/25/33 and every 12 weeks after (up to 2 years)
  ORR: the proportion of patients with confirmed complete response (CR) or partial response (PR), assessed by the independent review committee (IRC) according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.
Duration of response (DoR) | Week9/17/25/33 and every 12 weeks after (up to 2 years)
  DoR: the duration from the first evaluation as CR or PR to the first evaluation as progressive disease (PD) or death of any cause, per RECIST v1.1 assessed by investigator (INV) and IRC.
Disease control rate (DCR) | Week9/17/25/33 and every 12 weeks after (up to 2 years)
  DCR: the proportion of patients whose overall response is confirmed to be CR or PR or stable disease (SD) per RECIST v1.1, assessed by INV and IRC.
Investigator evaluated ORR | Week9/17/25/33 and every 12 weeks after (up to 2 years)
  the proportion of patients with confirmed CR or PR assessed by INV according to RECIST v1.1
Progression-free survival (PFS) | Week9/17/25/33 and every 12 weeks after (up to 2 years)
  the duration from the first date of treatment to the date of progression or death due to any cause, assessed by INV and IRC
Overall survival (OS) | from the first date of Infigratinib treatment until date of death.
  from the first date of Infigratinib treatment until date of death.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Center, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Second Hospital Lanzhou University, Lanzhou, Gansu
  - Dongguan City People's Hospital, Dongguan, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shandong Provincial Cancer Hosptial, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang